CLINICAL TRIAL: NCT03401307
Title: Central and Peripheral Nervous System Changes as Markers of Disease Progression in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Sepehr Mamoei, M.D., Ph.D.-Fellow, University of Southern Denmark
Other Study IDs: SDUSF-2016-106 - (660)
Record Dates: First submitted 2018-01-04; First posted 2018-01-17 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis; Neurodegeneration; Central Nervous System Lesion; Peripheral Nervous System Problem; Neurologic Deficits; Drug Effect; Genetic Disease; Neurophysiologic Abnormality
MeSH Terms: conditions — Multiple Sclerosis; Nerve Degeneration; Neurologic Manifestations; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples from blood for gene testing of the SORCS-3 gene.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders to Fampridine Treatment: Participants, who are classified as responders to Fampridine treatment, have already been identified in the MS-centers in the Region of Southern Denmark, where they undergo outpatient treatment and clinical controls. A 2-week Fampridine treatment phase, as described in the trial outline section, has been used to identify responders to Fampridine. Participants who improve with ≥20% on the T25FW are categorized as responders.
- Non-Responders to Fampridine Treatment: Participants, who are classified as non-responders to Fampridine treatment, have already been identified in the MS-centers in the Region of Southern Denmark, where they undergo outpatient treatment and clinical controls. A 2-week Fampridine treatment phase, as described in the trial outline section, has been used to identify non-responders to Fampridine. Participants who do not improve with ≥20% on the T25FW are categorized as non-responders.

SUMMARY:
OBJECTIVE To investigate neurodegeneration and demyelination in the central and peripheral nervous system in multiple sclerosis linked to disease progression and mechanisms that can explain different responses to Fampridine treatment in MS patients with walking disability.

METHOD The study is a prospective cohort follow-up study with 98 participants with MS and walking disability. Participants are identified as responders or non-responders to Fampridine treatment prior to the study. Participants will undergo MRI of the cerebrum with lesion load quantification, neurophysiological tests comprised of motor evoked potentials and electroneurographic examination, blood samples examining KIR4.1 antibodies, brain derived neurotrophic factor (BDNF), myelin protein zero (MPZ), peripheral myelin protein 22 (PMP22), p75-nerve growth factor receptor (p75NGFR) and anti-myelin associated glycoprotein (anti-MAG). The presence of SORCS-3 gene mutation will also be examined, as will cerebrospinal fluid levels of myelin basic protein, neurofilament heavy and light chains. Functional test of Timed 25-foot walk test (T25FW) will identify response to Fampridine treatment. A functional test battery will further detail function of upper extremities and cognition.

CONCLUSION This study will add to the understanding of neurodegeneration and demyelination in CNS and PNS in patients with MS having walking disability. This will impact clinical decision-making by improving organization of immunomodulatory treatment, identifying biomarkers thus facilitating earlier treatment and improving patient control, information and education.

DETAILED DESCRIPTION:
BACKGROUND Multiple Sclerosis (MS) is an autoimmune, inflammatory demyelinating disease targeting myelinated axons in the Central Nervous System (CNS). It is the most common nontraumatic cause of disability in young people. Most MS patients are diagnosed between the ages of 20 and 40 years. Denmark has a prevalence of approximately 155 MS patients per 100,000 inhabitants, which is among the highest in the world. The etiology of MS is not known, however, a combination of genetic and environmental factors is likely to be involved in triggering the disease.

CLINICAL PRESENTATION MS damages the CNS and causes progressive disability. Clinical symptoms of the patient depend on the location of the lesions that can occur anywhere in the CNS. Consequently the neurological impairments are very variable and consist of sensory, motor, visual, urinary, coordination and cognitive deficits. MS is divided into several categories based on disease progression: relapse-remitting multiple sclerosis (RRMS), secondary progressive multiple sclerosis (SPMS) and primary progressive multiple sclerosis (PPMS). Clinically isolated syndrome (CIS) is a single relapse compatible with MS accompanied by paraclinical evidence of demyelination with more than 80 percent of patients with CIS developing MS at a later stage.

WORKUP

McDonald criteria are used for diagnosing MS. They are based on clinical findings supported by paraclinical tests mentioned below. The aim is to demonstrate neurological impairments disseminated in time (lesions in the CNS are of different age) and localization in the CNS, while excluding other conditions:

1. Magnetic Resonance Imaging (MRI) of the brain and spinal cord is used to demonstrate lesions in the CNS.
2. Lumbar puncture is performed in order to demonstrate inflammation in the CNS. Analysis of the CSF can also exclude infection in the CNS.
3. Blood Samples are drawn to assess IgG, glucose and albumin in order to assess levels on both sides of the blood brain barrier (BBB) and to exclude other conditions.
4. Evoked Potentials are useful at identifying subclinical lesions.

   * Visual Evoked Potentials (VEP) assess the anterior visual pathways where delays in latencies indicates demyelination.
   * Somatosensory Evoked Potentials (SSEP) assess the posterior column of the spinal cord, brainstem and somatosensory cortex.

OTHER ASPECTS OF CURRENT WORKUP

The other aspects of the workup that are mentioned below, are not a part of the established workup on diagnosing or monitoring MS:

Blood Samples: Currently, there are no established peripheral blood biomarkers for MS. A study has demonstrated the SORCS3-gene as a potential MS risk gene. It has not been evaluated as a peripheral blood biomarker for MS as of yet, despite being potentially important in the pathogenesis of MS.

Furthermore a study has screened serum samples aiming to identify CNS-specific antibodies in MS.

Antibodies to the glial potassium channel KIR4.1 (Inward-rectifier potassium ion channel) was present in a subgroup of MS patients while being absent among patients with other neurological conditions and healthy controls.

Brain Derived Neurotrophic Factor (BDNF) is suggested to play a neuroprotective role in MS. BDNF concentrations has been shown to be lower in patients with RRMS compared to healthy controls.

There are currently biomarkers being indicative of demyelination in the PNS. Myelin protein zero (MPZ) is a cell surface component of myelin, which decreases in the tissue when demyelination occurs in the PNS. Peripheral myelin protein 22 (PMP22) is a glycoprotein component of myelin only found in the PNS, where it accounts for 2-5% of the myelin protein content.

The P75 nerve growth factor receptor (p75 NGFR) also known as P75 neurotrophin receptor (p75NTR) or low-affinity nerve growth factor receptor (LNGFR) is a ligand, which plays a role in Schwann cell migration and myelination during development, apoptosis and axonal regeneration. Anti-myelin associated glycoprotein (Anti-MAG) is a myelin marker that is rather specific for the PNS.

Neurophysiological tests: Motor Evoked Potentials (MEP) assess the motor pathways by stimulating the precentral gyrus. It is valuable in evaluating descending motor pathways, PNS and muscles. Electroneurographic examination (ENG) assesses the nerve conduction speed in the PNS and is not usually applied for patients with MS. Few studies that have evaluated examining nerve conduction speeds in the PNS among MS patients show that deficits in the PNS may be common among MS patients.

TREATMENT

There are three aspects of MS-treatment:

1. Immunomodulatory treatment with the aim of reducing/preventing relapses and slowing disease progression. Patients who are initiated in immunomodulatory treatment can be classified into two groups: responders or non-responders. The former profits from treatment while the latter does not respond or has marginal response to treatment. Responders can become non-responders after a while. Currently, the aim of immunomodulatory treatment among MS patients with RRMS, is no evidence of disease activity (NEDA), where the patient has no relapses, no increase in disability and no new active lesions on MRI.
2. Symptomatic treatment of walking disabilities, urinary tract problems, pain, depression, sexual problems, spasticity and fatigue. Neurorehabilitation is also an important part of the symptomatic treatment.
3. Treatment of relapses using high dose corticosteroids.

FAMPRIDINE Fampridine (Ampyra/Dalfampridine/4-aminopyridine) is the first oral agent approved by the Food and Drug Administration (FDA) and European Medicines Agency (EMA) for the treatment of walking disability in MS. It was approved in 2011 in Denmark for treatment of MS patients with walking disability.

Fampridine is a potassiumchannel blocker with a primary mechanism of action of blocking voltage-gated potassium channels. It blocks potassium from entering the channel, which leads to smoother nerve conduction and a subsequent improved amplitude and duration of the action potential. Fampridine acts at both the CNS and PNS and enhances nerve conduction in demyelinated axons and improves walking ability in a subset of MS patients. Furthermore a study has demonstrated improvement in cognition and upper extremity functioning, as a result of Fampridine treatment. Patients who do not profit from Fampridine treatment, are classified as non-responders. Currently, the mechanism behind non-response to Fampridine and conversion from response to non-response has not been studied. The functional test of T25FW is widely used to discriminate patients as responders or non-responders as well as to monitor response to treatment with Fampridine. When Fampridine treatment is indicated, patients will undergo a short-term treatment period while undergoing the T25FW in order to establish if there is response to treatment or non-response. If patients are classified as the latter, treatment will be stopped. During long-term treatment with Fampridine, the initial responders are yearly evaluated as to whether they are continuous responders.

SUMMARY OF STUDY RATIONALE Walking impairment is one of the most common symptoms of MS and has been reported as one of the most impactful symptoms on quality of life. MS patients with walking impairments receive the potassium-channel blocker, Fampridine, if they respond to this treatment. It has been established that approximately 35% of MS patients with walking disabilities are responders to this treatment, and thus have improvements in their walking speed and acceleration. The response status is established using the functional test T25FW. The presence of a specific potassiumchannel antibody (KIR 4.1) has been demonstrated in a subtype of MS patients while being absent in healthy controls. Antibodies affecting the PNS and thus aggravating walking abilities have been studied, but their links to MS remain to be investigated.

MS patients undergo neurodegeneration in the CNS with progressive neurological disability associated with axonal and neuronal damage, which is a major contributor to walking impairment. The involvement of the PNS in the dysfunction of the lower extremities as well as the role of the PNS as a potential marker of disease progression in MS remains to be fully elucidated. The effect of Fampridine in relation to the PNS has also not been examined and the mechanism behind non-response to Fampridine treatment and conversion from response to non-response remains to be elucidated.

Consequently, the overall research question of the present study proposal is to further clarify disease mechanisms involved in MS. Moreover, the overall aim of this project is to expand the knowledge on 1) neurodegeneration and demyelination in the central and peripheral nervous system in MS linked to disease progression over time and 2) to examine mechanisms that can explain the different responses to Fampridine treatment. Below, the specific study aims and hypotheses are outlined.

STUDY AIMS

Overall one main study is conducted, which has three inherent sub-studies. The aims of the main study Central and Peripheral Nervous System Changes as Markers of Disease Progression in Multiple Sclerosis are therefore:

1. to investigate the progression-rate and the corresponding changes, in patients with MS undertaking Fampridine treatment, in regards to a) magnetic resonance imaging-verified lesions in the central nervous system and b) neurophysiologic examinations of the peripheral nervous system. (Study I).
2. to investigate the response of potential peripheral blood biomarkers to Fampridine treatment in patients with MS. (Study II).
3. to compare motor pathways in the central nervous system and peripheral nervous system in patients with MS who are responders to non-responders of Fampridine treatment.

Null hypotheses are:

* Over time, among MS patients, there is neurodegeneration in the central nervous system while there is no neurodegeneration in the peripheral nervous system.
* There is no difference in biomarkers of the CNS and the PNS in MS patients.
* There are no differences in the motor pathways of the central and peripheral nervous system in patients with MS who respond and do not respond to treatment with Fampridine.
* Responders to Fampridine treatment do not convert to non-responders over time.

Participants will undergo MRI, blood samples, neurophysiologic examinations and the functional testing, as described in the trial outline section, in order to evaluate response to treatment with Fampridine and markers of disease progression. In addition to the widely used T25FW, additional functional tests will also be performed to have a more detailed overview of the function of the lower and upper extremities while also examining cognition over time. The T25FW test will also be used for identification of responders to treatment with Fampridine.

ELIGIBILITY:
Inclusion Criteria:

* Participants are diagnosed with MS according to the McDonald criteria.
* Categorized as responder or non-responder to Fampridine treatment.
* Age in the range of 18-65 years.
* Extended Disability Status Scale (EDSS) 4-7 points.
* Pyramidal Functions Score ≥ 2 in the Kurtzke Functional Systems Scores (FSS).

Exclusion Criteria:

* MS-attack and/or change in immunomodulatory treatment within 60 days before inclusion.
* Simultaneous use of medications that inhibit the organic cation transporter (OCT2).
* History of epileptic seizures.
* Clinically manifest heart-, liver-, kidney- (glomerular filtration rate < 80 ml/min), pulmonary disease, diabetes, alcohol intake exceeding the National Institute of Health's recommendations and pregnancy.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants in this cohort will be recruited from the four Multiple Sclerosis Centers in the Region of Southern Denmark (Sønderborg, Odense, Vejle/Kolding and Esbjerg), which (as of January 2016) have approximately 3600 patients with MS.
  Participants, who are classified as responders to Fampridine treatment, have already been identified in the MS-centers in the Region of Southern Denmark, where they undergo outpatient treatment and clinical controls. A 2-week Fampridine treatment phase, as described in the trial outline section, has been used to identify responders to Fampridine. Participants who improve with ≥20% on the T25FW are categorized as responders.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Timed 25-Foot Walk Test (T25FW) | Baseline up to 6, 12 and 18 months.
  The patient walks 25 feet as fast as possible. The test is repeated twice and the mean is used as the test result. This functional test measures walking speed and acceleration. This functional test has a high inter-rater and test-retest reliability and shows evidence of good concurrent validity. Hobart et al. have estimated the MCID for T25FW as an improvement >20% and Jensen et al. have recently estimated it to 17.8% when based on data distribution approach.

SECONDARY OUTCOMES:
Twelve Item MS Walking Scale (MSWS-12) | Baseline up to 6, 12 and 18 months.
  Questionnaire regarding assessment of walking speed from the perspective of the patient.
Guys Neurological Disability Scale (GNDS) | Baseline up to 6, 12 and 18 months.
  The Guy's Neurological Disability Scale (GNDS) is a clinical disability scale which encompass disabilities seen in multiple sclerosis. It has 12 separate categories which include cognition, mood, vision, speech, swallowing, upper limb function, lower limb function, bladder function, bowel function, sexual function, fatigue, and 'others'.
5-Times-Sit-to-Stand Test (5-STS) | Baseline up to 6, 12 and 18 months.
  The patient sits on a chair and stands up as fast as possible. This is repeated 5 times. Time stops when the patient has sat down up for the 5th time. This functional test measures strength and balance in lower extremities. The 5-STS shows validity and good test-retest and interobserver reliability. A 25.5% improvement on the 5-STS has been suggested to indicate true change and Jensen et al. have estimated the MCID to be 34.6%.
The Six Spot Step Test (SSST) | Baseline up to 6, 12 and 18 months.
  The patient walks in a crisscross pattern to six wooden markings on the floor as fast as possible while kicking each wooden disc to the side. The test is repeated twice with each leg and the mean is used as the test result. This functional test measures coordination, acceleration, speed and balancing. The re-test reliability and measurement error of the SSST is equally good as the T25FW. However, the sensitivity and discriminatory power of the SSST is better than that of the T25FW. Jensen et al. have estimated an MCID of 16.7%.
Antibodies | Baseline up to 12 months.
  Blood samples will be taken examining blood levels of KIR4.1 antibodies, brain derived neurotrophic factor (BDNF), myelin protein zero (MPZ), peripheral myelin protein 22 (PMP22), p75-nerve growth factor receptor (p75NGFR) and anti-myelin associated glycoprotein (anti-MAG). The aforementioned are know to have a role in (de)myelination in the PNS.
9-Hole Peg Test (9-HPT) | Baseline up to 6, 12 and 18 months.
  The patient undergoes this test with the dominant upper extremity and afterwards by the non-dominant upper extremity. 9 small pegs are placed into 9 holes and are removed and placed in a bowl as fast as possible. Time stops when the last peg is removed from the hole. The test is repeated twice for each upper limb and the mean is used as the test result for each upper limb. This functional test measures coordination and fine motor skills in the upper extremities. This test has high test-retest reliability. Jensen et al. have estimated an MCID of 15.3%.
Symbol Digit Modalities Test (SDMT) | Baseline up to 6, 12 and 18 months.
  The patient is presented to nine symbols, each representing a number from 0-9. A sheet containing 100 symbols should be paired with the corresponding numbers as fast as possible in 90 seconds. The amount of correct answers is the test result. This functional test measures cognition and more specifically processing speed. SDMT is sensitive for the detection of cognitive deterioration over time and is a reliable test over multiple test-retest intervals. Blum et al. have estimated the MCID for the SDMT as 5.1 arbitrary units (a.u.) and Jensen et al. have estimated an MCID as 17.1% and 6.2 a.u..
MRI of the brain | Baseline up to 12 months.
  MRI with T2-weighted sequences of the brain will be used to estimate the lesion load in the CNS, which will be compared to the clinical neurologic symptoms while serving as a reference to the MRI a year after. The locations of the T2 lesions and lesion load in the CNS will be compared between responders and non-responders to Fampridine treatment.
Neurophysiologic examinations | Baseline up to 12 months.
  MEP, combined with ENG, will be performed in order to investigate nerve conduction in the motor pathways of the CNS and PNS.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology (Skleroseklinikken), Sygehus Sønderjylland, Sønderborg, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mamoei S, Jensen HB, Pedersen AK, Nygaard MKE, Eskildsen SF, Dalgas U, Stenager E. Clinical, Neurophysiological, and MRI Markers of Fampridine Responsiveness in Multiple Sclerosis-An Explorative Study. Front Neurol. 2021 Oct 26;12:758710. doi: 10.3389/fneur.2021.758710. eCollection 2021. PMID 34764932
- [Derived] Mamoei S, Jensen HB, Dalgas U, Zijdewind I, Pedersen AK, Nygaard MKE, Eskildsen SF, Stenager E. A cross-sectional comparison of performance, neurophysiological and MRI outcomes of responders and non-responders to fampridine treatment in multiple sclerosis - An explorative study. J Clin Neurosci. 2020 Dec;82(Pt A):179-185. doi: 10.1016/j.jocn.2020.10.034. Epub 2020 Nov 15. PMID 33317729